CLINICAL TRIAL: NCT05824247
Title: A Prospective Cohort Study of 68ga-FAPI-pet-ct Versus FDG-pet-ct for Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: XMYY-2019-XJS1130
Record Dates: First submitted 2023-04-03; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; FAPI; PET-CT
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 68Ga-FAPI-PET-CT — a new technology that using Fibroblast activation protein （FAP）inhibitor as the tracer of PET-CT

SUMMARY:
A study to discuss the advantage of Fapi PET- CT in the initial diagnosis staging and lesion determination of ovarian cancer,whether it can be a evaluation strategy as an R0 evaluation tool or a prediction tool of chemotherapy response and evaluation of prognosis.

DETAILED DESCRIPTION:
Ovarian cancer is a challenging disease. It is difficult to diagnose early, and the recurrence rate is high after initial treatment. In the past decades, in addition to cancer treatment methods, imaging evaluation has also made corresponding progress. In particular, molecular imaging using FDG-PET / CT has shown a strong role in ovarian cancer. It can locate metabolic changes before anatomical changes, point out small lymph node (LN) metastasis, find distant metastasis and definite recurrence.In terms of diagnosis, several studies have shown that PET-CT is superior to CT in ovarian cancer staging and has obvious advantages in the determination of extraperitoneal metastasis; In terms of predicting whether ro surgery can be performed, there are some mature scoring systems, such as eisenkop,suidan score etc.but there is still no unique scoring mode suitable for PET-CT; Despite the above advantages, the nonspecific uptake mechanism of FDG-PET may lead to false positive results.Cancer associated fibroblasts (CAFs) are one of the factors that independently mediate tumor growth and metastasis. They are also related to extracellular fibrous tissue and tumor size Fibroblast activation protein (FAP) is overexpressed in fibroblasts of many epithelial cancers, but rarely expressed in normal tissues.Therefore, imaging with FAP as a marker is a promising way in many tumor types In our previous study, [68Ga] GA dotafapi - PET / CT D compared with [18F] - FDG PET / CT has advantages in detecting primary and metastatic lesions of many tumors, especially peritoneal metastatic tumors, such as ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary epithelial ovarian cancer confirmed by clinical consideration or puncture
2. PET-CT was chose as the initial imaging evaluation tool.

Exclusion Criteria:

1. Patients with acute inflammation
2. Lacking of clinical data
3. Severe complications and PET-CT contraindications

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary epithelial ovarian cancer confirmed by clinical consideration or puncture
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
coincidence rate | 1 year
  The consistency between the lesions detected by PET CT and those detected during operation (based on pathology)

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China